CLINICAL TRIAL: NCT00359281
Title: A Phase II, Fixed-sequenced, Open- Label, Research Study to Assess Pharmacokinetic Drug Interactions of AEGR-733 on Lipid-lowering Therapies in Healthy Volunteers
Brief Title: Pharmacokinetic Drug Interactions of AEGR-733 on Lipid-lowering Agents
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aegerion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: AEGR-733-002; Aegerion 002 PK study
Record Dates: First submitted 2006-07-31; First posted 2006-08-02 (Estimated); Results first posted 2014-03-04 (Estimated); Last update posted 2018-02-23 (Actual); Status verified 2018-02

CONDITIONS: Healthy
Keywords: healthy volunteers
MeSH Terms: interventions — Atorvastatin; Simvastatin; Ezetimibe; Fenofibrate; Dextromethorphan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: atorvastatin — Atrovastatin 20 mg and AEGR-733 10 mg or 60 mg
Drug: simvastatin — Simvastatin 20 mg and AEGR-733 10 mg or 60 mg
Drug: ezetimibe — Ezetimibe 10 mg and AEGR-733 10 mg
Drug: fenofibrate — Micronized Fenofibrate 145 mg and AEGR-733 10 mg
Drug: dextromethorphan — Dextromethorphan 30 mg and AEGR-733 10 mg
Drug: Extended Release Niacin — 1000 mg ER niacin and AEGR-733 10 mg

SUMMARY:
This phase II, open-label research study was conducted in 129 healthy volunteers. Each subject will be given one initial oral dose of one of 7 FDA-approved medications (probe drugs), followed by a 7 day period where subjects receive the study medication AEGR-733 at 10 or 60 mg. On study day 8 subjects will receive the second oral dose of the same probe drug that was given on day 1 and a last dose of AEGR-733 (total of 7 doses).Subjects will return in 1 week for a final safety visit. Each FDA- approved probe drug will be given to ten (10) or fifteen (15) subjects.

Safety, pharmacokinetic and pharmacodynamic assessments will be performed.

DETAILED DESCRIPTION:
Objectives:

Primary: To evaluate the effects of low and high doses of AEGR-733 on the pharmacokinetics of 6 FDA-approved medications that are likely to be used in combination with AEGR-733 as assessed by:

• Pharmacokinetic parameters: Cmax, Tmax, T1/2, and AUC (area under the curve).

Secondary: To evaluate the safety of AEGR-733 in combination with other lipid lowering agents in healthy subject as assessed by:

* Changes in associated liver enzymes AST, ALT and, Alkaline Phosphatase, & Total Bilirubin.
* Changes in all reported adverse events.
* To evaluate the effects of AEGR-733 in combination with other lipid lowering agents on the following lipids and lipoproteins: TC, LDL-C, VLDL, TG, HDL-C, ApoB and ApoAI.

4.0 STUDY DESIGN AND RATIONALE

4.1 STUDY DESIGN This is a single-center, phase II, clinical trial consisting of a eight (8) day open-label phase to assess the pharmacokinetic drug interactions of AEGR-733 on 6 probe drugs in healthy volunteers, followed by a one week safety visit. 105 subjects will be enrolled into this fixed-sequenced research study. Eligible subjects based on the screening visit will come to the GCRC for an inpatient visit (25-36 hr depending on if they come in evening before study day 1 or morning of). On the morning of study day 1, subjects will be assigned to one of 6 probe drugs(A-H below) and will take one dose of this medication. Timed blood samples will be drawn just before the administration of the probe drug and during the following times after drug administration (1,2,3,4,5,6,8,10,12,18, and 24 hrs). Prior to discharge after the 24 h blood sample, subjects will take an oral dose of AEGR-733 at 10 mg or 60 mg. Subjects will be given a 5 day supply of AEGR-733 at 10 mg or 60 mg to be taken once daily in the morning for the next 5 days (through day 7). On study day 8, subjects will take a final dose of AEGR-733 at 10 mg or 60 mg (total doses= 7) simultaneously with the same probe drug they took on day 1. Timed blood samples will be drawn just before the administration of the probe drug and AEGR-733 as well as 1,2,3,4,5,6,8,10,12,18, and 24 hours after study drug administration. After the 24 hour blood sample, subjects will be discharged. 15 subjects who participate in this study will receive dextromethorphan as the probe drug, which requires urine collection for 8 hours post dose. Blood for pharmacokinetic samples will not be collected on these subjects. Subjects receiving dextromethorphan may leave after the 8 hour urine collection at visits 2 and 3 (referred to as the inpatient visits). All subjects will come back 1 week later for a final visit to check safety lab parameters including liver transaminases and total bilirubin. Subjects will be instructed to abstain from drinking any alcoholic beverages once screened until study completion. Subjects who are not willing to comply with these requests will not be enrolled.

The FDA-approved lipid-lowering therapies will include:

A) Atorvastatin, 20 mg (n=15)and AEGR-733 10 mg B) Ezetimibe, 10 mg (n=10)and AEGR-733 10 mg C) Simvastatin, 20 mg (n=15)and AEGR-733 10 mg D) Rosuvastatin, 20 mg (n=10)and AEGR-733 10 mg E) Micronized fenofibrate, 145 mg (n=10)and AEGR-733 10 mg F) Atorvastatin, 20 mg (n=15) and AEGR-733 60 mg G) Rosuvastatin, 20 mg (n=15) and AEGR-733 60 mg H) Dextromethorphan, 30 mg (n=15) and AEGR-733 60 mg I) Extended Release Niacin, 1000 mg (n=20) and AEGR-733 10 mg

ELIGIBILITY:
Inclusion Criteria:

Males and non-pregnant/non-lactating female subjects between the ages of 18 and 70 who are in good overall health.

To be eligible for enrollment in this study, patients must meet all of the following criteria:

1. Men and women between the ages of 18 and 70
2. Women of child-bearing potential, that is, women not surgically sterilized and between menarche and 1 year post menopause, must test negative for pregnancy at the time of enrollment based on a urine pregnancy test and agree to use a reliable method of non-medication birth control (for example, a reliable barrier method of birth control [diaphragms with contraceptive jelly; cervical caps with contraceptive jelly; condoms with contraceptive foam; intrauterine devices]; partner with vasectomy; or abstinence) during the study and for one month following the last dose of study drug.
3. Subjects must be in good overall health
4. Subjects must be able to comprehend and willing to provide a signed IRB approved Informed Consent Form.
5. Subjects must be willing to comply with all study-related procedures.

Exclusion Criteria:

1. Known atherosclerotic cardiovascular disease, including coronary disease, cerebrovascular disease, or peripheral vascular disease
2. History of diabetes mellitus or fasting glucose > 126 mg/dL at the screening visit.
3. History of a non-skin malignancy within the previous 5 years
4. Renal insufficiency as defined by creatinine > 1.3 mg/dl
5. Any major active rheumatologic, pulmonary, or dermatologic disease or inflammatory condition
6. History of hypertension
7. Known coagulopathy and /or elevated PT/PTT >1.5 x ULN
8. Oral history of HIV positive
9. Patients who have undergone any organ transplant
10. Known active fibrotic or cirrhotic disease; ALT or AST > 1.5x ULN
11. Any major surgery within the previous 3 months
12. Individuals who currently use tobacco products or have done so in the previous 30 days
13. History of drug abuse (< 3 years)
14. Regular use of alcoholic beverages (> 7 drinks/day)
15. Subjects who do not agree to abstain from consuming alcoholic beverages during the entire study duration.
16. Body mass index (BMI) > 30 kg/m2 or < 18.5 kg/m2
17. Participation in an investigational drug study within 6 weeks prior to the screening visit
18. Serious or unstable medical or psychological conditions that, in the opinion of the investigator, would compromise the subject's safety or successful participation in the study will be excluded.
19. Currently taking any prescription, including oral contraceptives, or OTC medication regularly that cannot be stopped for at least 30 days prior to enrollment until completion of the study
20. Regular consumers of grapefruit juice, or have taken any medications known to be metabolized by CYP 3A4 within 4 weeks prior to the screening visit (ie. SSRIs, anti-fungals, anti-biotics, etc)
21. History of myalgia with a statin or unknown hypersensitivity to any statin, zetia, AEGR-733, or fenofibrate.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2006-03; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marina Cuchel, MD, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was performed from 19 May 2006 to 20 November 2007 at 1 medical clinic within the United States.
Groups:
- Atorvastatin 20 mg + Lomitapide 10 mg: One dose oral Atorvastatin 20 mg, Lomitapide 10 mg once daily 6 days then one dose oral Atorvastatin 20 mg and Lomitapide 10 mg
- Simvastatin 20 mg + Lomitapide 10 mg: One dose oral Simvastatin 20 mg, Lomitapide 10 mg once daily 6 days then one dose oral Simvastatin 20 mg and Lomitapide 10 mg
- Ezetimibe 10 mg + Lomitapide 10 mg: One dose oral Ezetimibe 10 mg, Lomitapide 10 mg once daily 6 days then one dose oral Ezetimibe 10 mg and Lomitapide 10 mg
- Rosuvastatin 20 mg + Lomitapide 10 mg: One dose oral Rosuvastatin 20 mg, Lomitapide 10 mg once daily 6 days then one dose oral Rosuvastatin 20 mg and Lomitapide 10 mg
- Fenofibrate 145 mg + Lomitapide 10 mg: One dose oral micronized Fenofibrate 145 mg, Lomitapide 10 mg once daily 6 days then one dose oral micronized Fenofibrate 145 mg and Lomitapide 10 mg
- Atorvastatin 20 mg + Lomitapide 60 mg: One dose oral Atorvastatin 20 mg, Lomitapide 60 mg once daily 6 days then one dose oral Atorvastatin 20 mg and Lomitapide 60 mg
- Rosuvastatin 20 mg + Lomitapide 60 mg: One dose oral Rosuvastatin 20 mg, Lomitapide 60 mg once daily 6 days then one dose oral Rosuvastatin 20 mg and Lomitapide 60 mg
- Dextrometh-rophan 30 mg + Lomitapide 60 mg: One dose oral Dextrometh-rophan 30 mg, Lomitapide 60 mg once daily 6 days then one dose oral Dextrometh-rophan 30 mg and Lomitapide 60 mg
- ER Niacin 1000 mg + Lomitapide 10 mg: One dose oral ER Niacin 1000 mg, Lomitapide 60 mg once daily 6 days then one dose oral ER Niacin 1000 mg and Lomitapide 60 mg
Period: Overall Study
Arm/Group | Atorvastatin 20 mg + Lomitapide 10 mg | Simvastatin 20 mg + Lomitapide 10 mg | Ezetimibe 10 mg + Lomitapide 10 mg | Rosuvastatin 20 mg + Lomitapide 10 mg | Fenofibrate 145 mg + Lomitapide 10 mg | Atorvastatin 20 mg + Lomitapide 60 mg | Rosuvastatin 20 mg + Lomitapide 60 mg | Dextrometh-rophan 30 mg + Lomitapide 60 mg | ER Niacin 1000 mg + Lomitapide 10 mg
Started | 16 | 15 | 10 | 10 | 10 | 15 | 18 | 15 | 20
Completed | 15 | 15 | 10 | 10 | 10 | 15 | 16 | 15 | 20
Not Completed | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Atorvastatin 20 mg + Lomitapide 10 mg | Simvastatin 20 mg + Lomitapide 10 mg | Ezetimibe 10 mg + Lomitapide 10 mg | Rosuvastatin 20 mg + Lomitapide 10 mg | Fenofibrate 145 mg + Lomitapide 10 mg | Atorvastatin 20 mg + Lomitapide 60 mg | Rosuvastatin 20 mg + Lomitapide 60 mg | Dextrometh-rophan 30 mg + Lomitapide 60 mg | ER Niacin 1000 mg + Lomitapide 10 mg | Total
Number analyzed (Participants) | 16 | 15 | 10 | 10 | 10 | 15 | 18 | 15 | 20 | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 26 (7) | 29 (12) | 29 (9) | 31 (13) | 24 (3) | 27 (8) | 31 (13) | 27 (9) | 29 (11) | 28 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 10 | 3 | 2 | 2 | 5 | 9 | 6 | 9 | 53
  Male | 9 | 5 | 7 | 8 | 8 | 10 | 9 | 9 | 11 | 76
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 2 | 0 | 0 | 1 | 3 | 1 | 3 | 2 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 1 | 4 | 2 | 1 | 5 | 2 | 4 | 23
  White | 11 | 11 | 8 | 5 | 7 | 6 | 11 | 10 | 13 | 82
  More than one race | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 0 | 5 | 1 | 0 | 1 | 8
Region of Enrollment [Number; unit: participants]
  United States | 16 | 15 | 10 | 10 | 10 | 15 | 18 | 15 | 20 | 129

OUTCOME MEASURES:

1. Primary Outcome: Area Under Concentration-time Curve From 0 to Last Measureable Concentration (AUC0-t) Atorvastatin Acid (Lomitapide 10 mg)
Description: Geometric Mean Ratio ln(AUC0-t) Day 8/Day 1 for atorvastatin acid (Lomitapide 10 mg)
Time Frame: 0 to 24 hour
Population: Pharmacokinetic
Measure: Geometric Mean (90% Confidence Interval); unit: Ratio
Arm/Group | Atorvastatin 20 mg + Lomitapide 10 mg
Number analyzed (Participants) | 15
Ratio | 110.97 [98.42 to 125.12]

2. Secondary Outcome: Percent Change From Baseline in Low-density Lipoprotein Cholesterol (LDL-C)
Description: Percent change from Baseline in LDL-C
Time Frame: Baseline to Day 8
Population: Intention To Treat
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Atorvastatin 20 mg + Lomitapide 10 mg | Simvastatin 20 mg + Lomitapide 10 mg | Ezetimibe 10 mg + Lomitapide 10 mg | Rosuvastatin 20 mg + Lomitapide 10 mg | Fenofibrate 145 mg + Lomitapide 10 mg | Atorvastatin 20 mg + Lomitapide 60 mg | Rosuvastatin 20 mg + Lomitapide 60 mg | Dextrometh-rophan 30 mg + Lomitapide 60 mg | ER Niacin 1000 mg + Lomitapide 10 mg
Number analyzed (Participants) | 16 | 15 | 10 | 10 | 10 | 15 | 18 | 15 | 20
Percent Change | -30.99 (14.47) | -26.43 (17.77) | -28.36 (12.53) | -41.74 (10.37) | -20.12 (25.56) | -66.02 (15.18) | -63.20 (18.59) | -46.07 (33.12) | -20.89 (15.17)

3. Primary Outcome: AUC0-t Simvastatin
Description: Geometric Mean Ratio ln(AUC0-t) Day 8/Day 1 for simvastatin
Time Frame: 0 to 24 hours
Population: Pharmacokinetic
Measure: Geometric Mean (90% Confidence Interval); unit: Ratio
Arm/Group | Simvastatin 20 mg + Lomitapide 10 mg
Number analyzed (Participants) | 15
Ratio | 162.25 [143.19 to 183.86]

4. Primary Outcome: AUC0-t Simvastatin Acid
Description: Geometric Mean Ratio ln(AUC0-t) Day 8/Day 1 for simvastatin acid
Time Frame: 0 to 24 hours
Population: Pharmacokinetic
Measure: Geometric Mean (90% Confidence Interval); unit: Ratio
Arm/Group | Simvastatin 20 mg + Lomitapide 10 mg
Number analyzed (Participants) | 15
Ratio | 138.76 [109.65 to 175.61]

5. Primary Outcome: AUC0-t Total Ezetimibe
Description: Geometric Mean Ratio ln(AUC0-t) Day 8/Day 1 for total ezetimibe
Time Frame: 0 to 24 hours
Population: Pharmacokinetic
Measure: Geometric Mean (90% Confidence Interval); unit: Ratio
Arm/Group | Ezetimibe 10 mg + Lomitapide 10 mg
Number analyzed (Participants) | 10
Ratio | 105.71 [92.62 to 120.66]

6. Primary Outcome: AUC0-t Rosuvastatin (Lomitapide 10 mg)
Description: Geometric Mean Ratio ln(AUC0-t) Day 8/Day 1 for rosuvastatin (Lomitapide 10 mg)
Time Frame: 0 to 24 hours
Population: Pharmacokinetic
Measure: Geometric Mean (90% Confidence Interval); unit: Ratio
Arm/Group | Rosuvastatin 20 mg + Lomitapide 10 mg
Number analyzed (Participants) | 10
Ratio | 102.05 [86.00 to 121.10]

7. Primary Outcome: AUC0-t Fenofibric Acid
Description: Geometric Mean Ratio ln(AUC0-t) Day 8/Day 1 for fenofibric acid
Time Frame: 0 to 24 hours
Population: Pharmacokinetic
Measure: Geometric Mean (90% Confidence Interval); unit: Ratio
Arm/Group | Fenofibrate 145 mg + Lomitapide 10 mg
Number analyzed (Participants) | 10
Ratio | 89.62 [82.76 to 97.04]

8. Primary Outcome: AUC0-t Atorvastatin Acid (Lomitapide 60 mg)
Description: Geometric Mean Ratio ln(AUC0-t) Day 8/Day 1 for atorvastatin acid (Lomitapide 60 mg)
Time Frame: 0 to 24 hours
Population: Pharmacokinetic
Measure: Geometric Mean (90% Confidence Interval); unit: Ratio
Arm/Group | Atorvastatin 20 mg + Lomitapide 60 mg
Number analyzed (Participants) | 15
Ratio | 152.32 [133.76 to 173.45]

9. Primary Outcome: AUC0-t Rosuvastatin (Lomitapide 60 mg)
Description: Geometric Mean Ratio ln(AUC0-t) Day 8/Day 1 for rosuvastatin (Lomitapide 60 mg)
Time Frame: 0 to 24 hours
Population: Pharmacokinetic
Measure: Geometric Mean (90% Confidence Interval); unit: Ratio
Arm/Group | Rosuvastatin 20 mg + Lomitapide 60 mg
Number analyzed (Participants) | 15
Ratio | 132.21 [111.56 to 156.70]

10. Primary Outcome: AUC0-t Nicotinic Acid
Description: Geometric Mean Ratio ln(AUC0-t) Day 8/Day 1 for nicotinic acid
Time Frame: 0 to 24 hours
Population: Pharmacokinetic
Measure: Geometric Mean (90% Confidence Interval); unit: Ratio
Arm/Group | ER Niacin 1000 mg + Lomitapide 10 mg
Number analyzed (Participants) | 20
Ratio | 110.22 [78.28 to 155.18]

11. Primary Outcome: AUC0-t Nicotinuric Acid
Description: Geometric Mean Ratio ln(AUC0-t) Day 8/Day 1 for nicotinuric acid
Time Frame: 0 to 24 hours
Population: Pharmacokinetic
Measure: Geometric Mean (90% Confidence Interval); unit: Ratio
Arm/Group | ER Niacin 1000 mg + Lomitapide 10 mg
Number analyzed (Participants) | 20
Ratio | 79.15 [59.82 to 104.72]

ADVERSE EVENTS:
Time Frame: From the first dose of study drug (Day 1) to 14 days after the first dose (Day 15)
Arm/Group | Atorvastatin 20 mg + Lomitapide 10 mg | Simvastatin 20 mg + Lomitapide 10 mg | Ezetimibe 10 mg + Lomitapide 10 mg | Rosuvastatin 20 mg + Lomitapide 10 mg | Fenofibrate 145 mg + Lomitapide 10 mg | Atorvastatin 20 mg + Lomitapide 60 mg | Rosuvastatin 20 mg + Lomitapide 60 mg | Dextrometh-rophan 30 mg + Lomitapide 60 mg | ER Niacin 1000 mg + Lomitapide 10 mg
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/15 | 0/10 | 0/10 | 0/10 | 0/15 | 0/18 | 0/15 | 0/20
Other Adverse Events (participants affected / at risk) | 8/16 | 8/15 | 6/10 | 3/10 | 6/10 | 12/15 | 15/18 | 11/15 | 18/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Atorvastatin 20 mg + Lomitapide 10 mg (N=16) | Simvastatin 20 mg + Lomitapide 10 mg (N=15) | Ezetimibe 10 mg + Lomitapide 10 mg (N=10) | Rosuvastatin 20 mg + Lomitapide 10 mg (N=10) | Fenofibrate 145 mg + Lomitapide 10 mg (N=10) | Atorvastatin 20 mg + Lomitapide 60 mg (N=15) | Rosuvastatin 20 mg + Lomitapide 60 mg (N=18) | Dextrometh-rophan 30 mg + Lomitapide 60 mg (N=15) | ER Niacin 1000 mg + Lomitapide 10 mg (N=20)
Diarrhoea (Gastrointestinal disorders) | 3 | 4 | 1 | 0 | 3 | 7 | 9 | 4 | 2
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 2 | 2 | 3 | 3 | 2
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 5 | 2 | 5 | 1
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 12
Headache (Nervous system disorders) | 0 | 2 | 1 | 2 | 0 | 1 | 1 | 0 | 3
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 2 | 1 | 2
Abnormal faeces (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 3
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 4
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 7
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 3 | 1 | 0 | 0 | 1 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 2
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eructation (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chromaturia (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Faeces hard (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infusion site haematoma (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastric dilatation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infusion site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other